CLINICAL TRIAL: NCT02664376
Title: Prevalence of Sarcopenia and Its Geriatric Features
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Murielle Surquin, Head of clinic, Brugmann University Hospital
Other Study IDs: CHUB-sarcopenia
Record Dates: First submitted 2016-01-19; First posted 2016-01-27 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Sarcopenia
Keywords: sarcopenia; geriatry
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric ward population: Every patient aged over 65 admitted in the unit 83 of the Geriatry Department, CHU Brugmann Hospital, undergoes a global geriatric evaluation at the end of its hospitalisation stay, including sarcopenia detection.
  Interventions: Other: Sarcopenia detection

INTERVENTIONS:
Other: Sarcopenia detection — The assessment of sarcopenia is performed according to the recommendations of the EWGSOP (European Working Group on Sarcopenia in Older people). Three measurements are made:
  * Muscle mass measurement by dual energy X-ray absorptiometry (DEXA).
  * Walking speed measurement
  * Hand grip test
  A diagnosis of sarcopenia is established if the walking speed is inferior to 0.8 m/sec, the muscular strength is low and the muscular mass is low.
  Data regarding the geriatric characteristics of this sarcopenic population will be collected.

SUMMARY:
The goal of this study is to determine the prevalence of sarcopenia in a geriatric hospital ward.

Sarcopenia is defined by a loss of muscle mass, loss of muscle strength and loss of muscle quality. It is a geriatric syndrome that, to this date, is not systematically tracked in clinical practice.

In order to detect sarcopenia, the investigators will use the operational definition proposed by the European Working Group (EWGSOP) involving the measure of three parameters, namely the speed of walking, the muscle strength and the measurement of the muscular mass.

ELIGIBILITY:
Inclusion Criteria:

* To be admitted in the unit 83 of the Geriatric Departement of the CHU Brugmann hospital, from 10/01/2016 till 30/03/2017.

Exclusion Criteria:

* Patients unable to consent or without representatives
* Patients unable to perform the hand- grip test, the walk test or measurement of the body components by DEXA
* Patients in severe pain
* Bedridden patients
* Patients for which a clear therapeutic abstention has been established
* Language barriere that cannot be overcome
* Patients unable to walk without the help of a third person

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Each patient over 65 years admitted to the unit 83 of the Geriatric Department, CHU Brugmann Hospital, from 10/01/2016 till 30/03/2017 undergoes a comprehensive geriatric assessment at the end of its hospitalisation stay. The screening for sarcopenia is part of this geriatric assessment.
Sampling Method: Non-Probability Sample
Enrollment: 834 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Prevalence of sarcopenia | From 10/01/2016 till 30/03/2017 (up to 15 months)
  Sarcopenia detection will be performed at the end of each hospitalization stay in unit 83 of the CHU Brugmann Hospital (Geriatry Department)

SECONDARY OUTCOMES:
Percentage of hospitalized patients unable to perform the sarcopenia detection test | From 10/01/2016 till 30/03/2017 (up to 15 months)
  Systematic retrospective review of patients hospitalised in the geriatric ward of the CHU Brugmann hospital during the length of the study, in order to determine the percentage of patients that could not, because of one of more exclusion criteria, perform the sarcopenia detection test.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Barré, MD, Principal Investigator — CHU Brugmann; Murielle Surquin, MD, Principal Investigator — CHU Brugmann; Florence Benoît, MD, Principal Investigator — CHU Brugmann; Marie Claessens, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Baumgartner RN, Koehler KM, Gallagher D, Romero L, Heymsfield SB, Ross RR, Garry PJ, Lindeman RD. Epidemiology of sarcopenia among the elderly in New Mexico. Am J Epidemiol. 1998 Apr 15;147(8):755-63. doi: 10.1093/oxfordjournals.aje.a009520. PMID 9554417
- [Background] Cesari M, Kritchevsky SB, Newman AB, Simonsick EM, Harris TB, Penninx BW, Brach JS, Tylavsky FA, Satterfield S, Bauer DC, Rubin SM, Visser M, Pahor M; Health, Aging and Body Composition Study. Added value of physical performance measures in predicting adverse health-related events: results from the Health, Aging And Body Composition Study. J Am Geriatr Soc. 2009 Feb;57(2):251-9. doi: 10.1111/j.1532-5415.2008.02126.x. PMID 19207142
- [Background] Lauretani F, Russo CR, Bandinelli S, Bartali B, Cavazzini C, Di Iorio A, Corsi AM, Rantanen T, Guralnik JM, Ferrucci L. Age-associated changes in skeletal muscles and their effect on mobility: an operational diagnosis of sarcopenia. J Appl Physiol (1985). 2003 Nov;95(5):1851-60. doi: 10.1152/japplphysiol.00246.2003. PMID 14555665